CLINICAL TRIAL: NCT01884272
Title: A Phase 1 Study to Evaluate the Potential Two-Way Pharmacokinetic Interaction Between Lesinurad and Naproxen and Between Lesinurad and Indomethacin in Healthy Adult Male Subjects
Brief Title: NSAID Drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RDEA594-126
Record Dates: First submitted 2013-06-18; First posted 2013-06-24 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — lesinurad; Naproxen; Indomethacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lesinurad 400 mg and naproxen 250 mg (Experimental): Lesinurad once daily (qd) Day 1, naproxen twice daily (bid) Day 2-6, lesinurad qd with naproxen bid Day 7-14.
  Interventions: Drug: lesinurad 400 mg; Drug: naproxen 250 mg
- Lesinurad 400 mg and indomethacin 25 mg (Active Comparator): Lesinurad qd Day 1, indomethacin bid Day 2-6, lesinurad qd with indomethacin bid Day 7-14.
  Interventions: Drug: lesinurad 400 mg; Drug: indomethacin 25 mg

INTERVENTIONS:
Drug: lesinurad 400 mg
Drug: naproxen 250 mg
  Arms: Lesinurad 400 mg and naproxen 250 mg
Drug: indomethacin 25 mg
  Arms: Lesinurad 400 mg and indomethacin 25 mg

SUMMARY:
This is a drug-drug interaction study in healthy volunteers to evaluate the potential pharmacokinetic (PK) effects of non-steroidal anti-inflammatory drugs on lesinurad and leinurad on the non-steroidal anti-inflammatory drugs.

DETAILED DESCRIPTION:
Naproxen and indomethacin are non-steroidal anti-inflammatory drugs (NSAIDs) used both prophylactically for the prevention of, and as a treatment for, acute gout flares. RDEA594-126 is an open-label study designed to assess the potential effect of multiple doses of naproxen and indomethacin on the single-dose PK of lesinurad, and to assess the potential effect of multiple doses of lesinurad on the multiple-dose PK of naproxen and indomethacin.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body weight ≥ 50 kg (110 lbs) and a body mass index (BMI) ≥ 18 and ≤ 30 kg/m2.
* Subject is free of any clinically significant disease that requires a physician's care and/or would interfere with study evaluations or procedures.
* Subject has no clinically relevant abnormalities in vital signs, ECG, physical examination or safety laboratory values.

Exclusion Criteria:

* Subject has clinically significant pulmonary, cardiovascular, gastrointestinal, neurologic, hepatic, renal, urological, or psychiatric disorders.
* Subject has a history or suspicion of kidney stones.
* Subject has a history of asthma.
* Subject has undergone major surgery within 3 months prior to Day 1.
* Subject has donated blood or experienced significant blood loss (> 450 mL) within 12 weeks prior to Day 1 or gave a plasma donation within 4 weeks prior to the Screening visit.
* Subject has inadequate venous access or unsuitable veins for repeated venipuncture.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
PK profile of lesinurad from plasma and urine | Day 1, Day 6 (urine only), Day 7, Day 14
  Profile in terms of AUC, Tmax, Cmax, and t1/2 AUC: area under the plasma concentration versus time curve; Tmax: time to maximum plasma concentration; Cmax: maximum plasma drug concentration; t1/2: apparent terminal half-life
PK profile of naproxen and indomethacin from plasma and urine | Day 1, Day 6 (urine only), Day 7, Day 14
  Profile in terms of AUC, Tmax, Cmax, and t1/2

SECONDARY OUTCOMES:
Incidence of Adverse Events and Changes in Laboratory, Electrocardiogram, and Vital Signs Parameters | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: S Bradley, MD, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Kalamazoo, Michigan, United States